CLINICAL TRIAL: NCT03354585
Title: Brain Mechanisms Supporting Mindfulness-based Chronic Pain Relief
Brief Title: Mindfulness and Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Fadel Zeidan, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 181814
Record Dates: First submitted 2017-10-16; First posted 2017-11-28 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Chronic Low Back Pain
Keywords: Mindfulness; fMRI; Pain; Low Back; Radicular
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This intervention study will utilize an unbiased randomized study design. Pain intensity and pain unpleasantness ratings will be assessed using before and after all sessions where low back pain is induced. Study volunteers will be randomized and subsequently participate in a six session mindfulness meditation, non-mindfulness meditation or book-listening control regimen. Study volunteers will be required to complete two MRI scans over the course of the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the study physician, research coordinator, and intervention facilitators will be aware of group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mindfulness group (Experimental): Study volunteers will participate in a six-session meditation training regimen. In brief, subjects will be taught that perceived sensory events are "momentary" and "fleeting" and do not require further evaluation. There will be an emphasis on breath focus and altering one's perspective of discursive sensory events. This intervention has been found to reliably attenuate the subjective experience of pain.
  Interventions: Behavioral: mindfulness training
- non-mindfulness group (Sham Comparator): Study volunteers will participate in a six-session meditation training regimen. In brief, subjects will be taught to take deep breaths and relax.
  Interventions: Behavioral: non-mindfulness training
- book-listening (Active Comparator): Study volunteers will listen to an audio recording of the Natural History of Selborne across each session.This 6 session intervention is meant to provide the control attention to the facilitator, room setting, social support, conditioning, and the time elapsed during the other respective interventions. We do not expect that this group will demonstrate significant cerebral blood flow changes as a function of the intervention.
  Interventions: Behavioral: book-listening

INTERVENTIONS:
Behavioral: mindfulness training — A well-validated brief mindfulness-based mental training regimen [20 min/session(s)] will be used to teach patients to independently practice mindfulness. Participants will be asked to close their eyes acknowledge distracting thoughts and feelings.
  Other Names: mental training
  Arms: mindfulness group
Behavioral: non-mindfulness training — A well-validated brief meditation-based mental training regimen [20 min/session(s)] will be used to teach patients to independently practice deep breathing. Participants will be asked to close their eyes acknowledge distracting thoughts and feelings.
  Other Names: mental training
  Arms: non-mindfulness group
Behavioral: book-listening — Study volunteers will listen to The Natural History and Antiquities of Selborne throughout the intervention.
  Arms: book-listening

SUMMARY:
The purpose of this study is to see if mindfulness, a form of mental training, or listening to a book alters brain activation in response to raising your leg that may produce the feeling of pain. A technique called functional magnetic resonance imaging (fMRI) allows scientists to determine which parts of the brain are active during a particular task. This study will provide new information about how mindfulness affects the brain.

DETAILED DESCRIPTION:
To determine if mindfulness meditation-induced reductions in chronic low back pain (cLBP) patients will be associated with greater anterior insula (aINS), orbitofrontal cortex (OFC), subgenual anterior cingulate cortex (sgACC), and/or thalamic deactivation when compared to rest, the sham-mindfulness meditation and the book-listening control groups. One-hundred and twenty individuals will be randomized to a mindfulness meditation (n=40), non-mindfulness meditation (n=40) and book-listening-control (n=40). Each participants will be administered noxious heat and the chronic low back pain evoking, straight leg raise test during fMRI.

ELIGIBILITY:
Inclusion criteria are:

* Participants must have a medical evaluation that demonstrates chronic low back pain that is evoked by lifting the legs. Existing medical records, per physician discretion and low back examinations will confirm diagnosis. This will be determined over the phone during the (pre) screening and at study session 1, and will not be contingent on MRI.
* Participants must be between the ages of 18-65 years.
* Participants must rate their daily chronic pain intensity at a 3 or greater on 0-10 visual analog scale.
* Participants must have experienced their radicular pain for at least 3 months duration.
* Participants must be right-handed.
* Participants must have no prior meditative experience

Exclusion criteria:

* Participants must not be participating in any new (within 2 weeks prior or anytime after enrollment) pain management procedures during the study period.
* Participants must not have had back surgery within the last year before their enrollment into the study.
* Participants must not have had any other sensory or motor deficits that precludes participation in this study.
* Participants must not have known anomalies of the central nervous system including: stroke, dementia, aneurysm, a personal history of psychosis.
* Participants must not have metal implants including ferrous arterial stints or coils, spinal stimulators, pacemakers, or defibrillators, permanently implanted hearing aides, bullets, BBs, or pellets, retinal eye implants, infusion pump for insulin or other medicines, ferrous surgical clips, staples, metal sutures, orthopedic hardware above or including the shoulders, body piercings that cannot be removed.
* Participants must not be claustrophobic.
* Participants must not produce negative straight leg test (i.e. a test is considered positive when the person reports reproducible pain at 40 degrees of hip flexion or less).
* Participants must not be pregnant
* Participants must not be over 275 pounds

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Cerebral Blood Flow (average blood perfusion; mL blood/100 grams tissue/minute) | There will be up to 2 fMRI sessions (Visit 2, and 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  Changes in cerebral blood flow will be assessed during pseudo continuous arterial spin labeling fMRI during their respective manipulations.

SECONDARY OUTCOMES:
Visual Analog Scale Pain Ratings | Baseline and 3 fMRI sessions (Visit 1, 2, 9, and 16). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  Changes in visual analog scale (VAS) pain ratings will be assessed in response to the straight leg raise test and lying supine in the MRI scanner.
  Psychophysical Assessment of Pain: As previously in all of our previous pain studies, pain intensity and unpleasantness ratings will be assessed with a Visual Analog Scale. These scales 1) provide reliably separate assessment of experimental and clinical pain intensity and unpleasantness, 2) are internally consistent, and 3) approximate ratio scale measurement accuracy. The minimum rating ("0") is designated as "no pain" whereas the maximum ("10") is labeled as "most intense imaginable" or "most unpleasant imaginable".
  Higher numbers correspond to higher perceived pain
Numerical Pain Ratings | Two fMRI sessions. Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  Changes in numerical pain ratings (NRS) will be assessed in response to the straight leg raise test and lying supine in the MRI scanner.
  Psychophysical Assessment of Pain: As previously in all of our previous pain studies, pain intensity and unpleasantness ratings will be assessed with a Visual Analog Scale. These scales 1) provide reliably separate assessment of experimental and clinical pain intensity and unpleasantness, 2) are internally consistent, and 3) approximate ratio scale measurement accuracy. The minimum rating ("0") is designated as "no pain" whereas the maximum ("10") is labeled as "most intense imaginable" or "most unpleasant imaginable".
  Higher numbers correspond to higher perceived pain
Blood Oxygen Dependent Signaling | Two fMRI sessions. Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  Changes in BOLD fMRIacquired during noxious heat stimulation during rest and manipulations Psychophysical Assessment of Pain: As previously in all of our previous pain studies, pain intensity and unpleasantness ratings will be assessed with a Visual Analog Scale. These scales 1) provide reliably separate assessment of experimental and clinical pain intensity and unpleasantness, 2) are internally consistent, and 3) approximate ratio scale measurement accuracy. The minimum rating ("0") is designated as "no pain" whereas the maximum ("10") is labeled as "most intense imaginable" or "most unpleasant imaginable".
  Higher numbers correspond to higher perceived pain
Respiration Rate | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  Respiration rate will be collected and recorded on a Biopac respiratory transducer. Changes in respiration rate could be predictive of analgesia and health promotion.
Five Facet Mindfulness Questionnaire | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a 39-item multidimensional measure of trait mindfulness and includes five subscales: non-reactivity, nonjudgment, describing, observing, and acting with awareness. A numeric value between 1 (never or very rarely true) and 5 (very often or always true) is provided in response to each statement.
PROMIS Pain Behavior Measure | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a 5-item questionnaire that measures complaints of suffering, verbal or nonverbal (i.e. such as when I am in pain I squirm) from the past 7 days. Scoring for this measure is item-content dependent.
Brief Pain Inventory | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is an 8-item assessment widely used to measure clinical pain. Higher scores reflect a higher severity rating of pain.
Pain Catastrophizing Scale | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a 13-item questionnaire with 3 subscales assessing rumination, magnification, and helplessness in patients. A numeric value between 0 (not at all) and 4 (all the time) is provided in response to each statement. Scores on this assessment range from 0 to 52, with higher values reflecting more salient impacts of pain on one's day to day experience.
Beck Depression Inventory | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a 21-item standard assessment used to measure clinical depression. Scores on this assessment range from 0 to 63, where higher scores indicate higher levels of depression.
Freiburg Mindfulness Inventory | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a 14-item standard mindfulness scale to measure potential changes in mindfulness before and after intervention. A rating between "rarely" (0) to "often" (4) is provided in response to each statement.
Roland-Morris Disability Questionnaire | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a critical assessment for assessing the functional impact of chronic low back pain. Scores on this assessment range from 0 to 24, where higher scores indicate greater disability and limited functioning due to pain.
Cohen Perceived Stress Scale | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  The CPS is a series of 10 temporally constrained (i.e. in the last month) questions meant to ascertain the relative frequency of stressors in one's life, ranging from never (scored as 0) to very often (scored as 4). All positively stated questions are reversed scored and then all items are summed to yield a final estimate of stress. The higher the score the higher the level of stress.

OTHER OUTCOMES:
Social Connectedness Scale | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a 20-item assessment designed to measure social connectedness, an attribute of the self that reflects cognitions of enduring interpersonal closeness with the social world, in participants. Higher scores on the Social Connectedness Scale reflect a stronger sense of social connectedness, there are no sub-scales. The minimum score is 20 and the maximum score is 120.
Perceived Intervention Effectiveness | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This measure will be assessed with a VAS ("0" = not effective at all; "10"= most effective imaginable) for each intervention session's respective manipulation.
Positive and Negative Affect Scale | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a 20-item self-report assessment used to assess positive and negative affect in a participant. A rating between "very slightly or not at all" (1) to "extremely" (5) is provided in response to each statement. Higher scores indicate a greater level of positive affect, and a lower score reveals a greater level of negative affect.
Pittsburgh Sleep Quality Index | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a 10-item assessment designed to measure quality of sleep. This measure is scored along a 5-point Likert scale with values ranging from 0 to 5, specific ratings associated with particular items. Scores on this assessment range from 0 to 28, with higher values reflecting greater levels of insomnia.
SF 12 Health Survey | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a 12-item version of the SF-36 item Health Survey designed to assess general mental and physical functioning, and overall health-related quality of life. Scores on this assessment range from 0 to 100, where a higher score indicates a higher level of overall health.
State Anxiety Inventory | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This inventory is a 20-item assessment used to measure a subject's state of anxiety. A numeric value between 1 (Not at all) and 4 (Very Much So) is provided in response to each statement. The range of scores for this test is between 20 and 80, with higher scores reflecting higher estimates of anxiety.
PROMIS Pain Quality Measure | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a 5-item questionnaire that measures sensory quality of pain experience (throbbing, aching, etc). A numeric value between 1 (not at all) and 5 (very much) is provided in response to each statement. Higher scores indicate a greater quality of pain.
PROMIS 29-Item Profile | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a 29-item generic health-related survey that assesses 7 domains with 4-items in each domain: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participant in social roles/activities. Higher scores represent different outcomes based on domain. Higher scores on symptom-oriented domains represent worse symptomatology, but higher scores on function-oriented domains represent better functioning.
Patients' Global Impression of Change | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a self-report assessment measured on a 7-point scaled designed to evaluate perceived improvement over trial/efficacy of treatment. Options range from "no change" to "a great deal better, and a considerable improvement that has made all the difference." Higher ratings indicate greater impressions of change.
Profile of Mood States Form | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a 40-item core measure of emotional functioning and includes 6 mood states: tension-anxiety, depression-dejection, anger-hostility, vigor-activity, fatigue-inertia, and confusion-bewilderment. A numeric value between 1 (not at all) and 5 (extremely) is provided in response to each statement. Total mood disturbance scoring is calculated by summing the totals for the negative subscales and then subtracting the totals for the positive subscales.
Pain Self Efficacy Questionnaire | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a 10-item questionnaire that's designed to assess the confidence in people with ongoing pain have in performing activities while in pain. The option of either "not at all confident" or "completely confident" is posed after each item. Scores on this assessment range from 0 to 60, with higher scores indicating stronger self-efficacy beliefs.
Chronic Pain Acceptance Questionnaire | There will be up to 2 fMRI sessions (Visit 2, 9). Active enrollment provides up to 8 weeks to complete all study interventions, scans, and assessments.
  This is a 20-item assessment designed to measure acceptance of pain. Items are rated on a 7-point scale from 0 (never true) to 6 (always true). Higher scores indicate higher levels of acceptance.

CONTACTS AND LOCATIONS:
Overall Officials: Fadel Zeidan, PhD, Principal Investigator — Principal Investigator
Locations (2):
- United States (2):
  - UC San Diego, La Jolla, California
  - UC San Diego Center for Functional MRI, La Jolla, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Apkarian AV, Krauss BR, Fredrickson BE, Szeverenyi NM. Imaging the pain of low back pain: functional magnetic resonance imaging in combination with monitoring subjective pain perception allows the study of clinical pain states. Neurosci Lett. 2001 Feb 16;299(1-2):57-60. doi: 10.1016/s0304-3940(01)01504-x. PMID 11166937
- [Background] Bruno PA, Millar DP, Goertzen DA. Inter-rater agreement, sensitivity, and specificity of the prone hip extension test and active straight leg raise test. Chiropr Man Therap. 2014 Jun 16;22:23. doi: 10.1186/2045-709X-22-23. eCollection 2014. PMID 24982755
- [Background] Chen X, Spaeth RB, Freeman SG, Scarborough DM, Hashmi JA, Wey HY, Egorova N, Vangel M, Mao J, Wasan AD, Edwards RR, Gollub RL, Kong J. The modulation effect of longitudinal acupuncture on resting state functional connectivity in knee osteoarthritis patients. Mol Pain. 2015 Oct 29;11:67. doi: 10.1186/s12990-015-0071-9. PMID 26511911
- [Background] Cropley M, Ussher M, Charitou E. Acute effects of a guided relaxation routine (body scan) on tobacco withdrawal symptoms and cravings in abstinent smokers. Addiction. 2007 Jun;102(6):989-93. doi: 10.1111/j.1360-0443.2007.01832.x. PMID 17523994
- [Background] Eisenach JC, Rauck RL, Curry R. Intrathecal, but not intravenous adenosine reduces allodynia in patients with neuropathic pain. Pain. 2003 Sep;105(1-2):65-70. doi: 10.1016/s0304-3959(03)00158-1. PMID 14499421
- [Background] Eisenach JC, Thomas JA, Rauck RL, Curry R, Li X. Cystatin C in cerebrospinal fluid is not a diagnostic test for pain in humans. Pain. 2004 Feb;107(3):207-212. doi: 10.1016/j.pain.2003.09.007. PMID 14736582
- [Background] Fardon DF. Nomenclature and classification of lumbar disc pathology. Spine (Phila Pa 1976). 2001 Mar 1;26(5):461-2. doi: 10.1097/00007632-200103010-00007. No abstract available. PMID 11242371
- [Background] Fardon DF, Williams AL, Dohring EJ, Murtagh FR, Gabriel Rothman SL, Sze GK. Lumbar disc nomenclature: version 2.0: Recommendations of the combined task forces of the North American Spine Society, the American Society of Spine Radiology and the American Society of Neuroradiology. Spine J. 2014 Nov 1;14(11):2525-45. doi: 10.1016/j.spinee.2014.04.022. Epub 2014 Apr 24. PMID 24768732
- [Background] Jamison RN, Ross EL, Michna E, Chen LQ, Holcomb C, Wasan AD. Substance misuse treatment for high-risk chronic pain patients on opioid therapy: a randomized trial. Pain. 2010 Sep;150(3):390-400. doi: 10.1016/j.pain.2010.02.033. Epub 2010 Mar 23. PMID 20334973
- [Background] Kwong EH, Virani N, Robert M, Gerry K, Harding A, Rose MS, Dukelow SP, Barton PM. Inter-rater reliability of the Active Straight-Leg Raise and One-Leg Standing tests in non-pregnant women. J Rehabil Med. 2013 Nov;45(10):1058-64. doi: 10.2340/16501977-1213. PMID 23995959
- [Background] Lazar N (2008) The Statistical Analysis of Functional MRI Data. New York, New York: Springer.
- [Background] Loggia ML, Kim J, Gollub RL, Vangel MG, Kirsch I, Kong J, Wasan AD, Napadow V. Default mode network connectivity encodes clinical pain: an arterial spin labeling study. Pain. 2013 Jan;154(1):24-33. doi: 10.1016/j.pain.2012.07.029. Epub 2012 Oct 27. PMID 23111164
- [Background] Mens JM, Vleeming A, Snijders CJ, Stam HJ, Ginai AZ. The active straight leg raising test and mobility of the pelvic joints. Eur Spine J. 1999;8(6):468-73. doi: 10.1007/s005860050206. PMID 10664304
- [Background] Pantano P, Mainero C, Lenzi D, Caramia F, Iannetti GD, Piattella MC, Pestalozza I, Di Legge S, Bozzao L, Pozzilli C. A longitudinal fMRI study on motor activity in patients with multiple sclerosis. Brain. 2005 Sep;128(Pt 9):2146-53. doi: 10.1093/brain/awh549. Epub 2005 May 18. PMID 15901646
- [Background] Quiton RL, Keaser ML, Zhuo J, Gullapalli RP, Greenspan JD. Intersession reliability of fMRI activation for heat pain and motor tasks. Neuroimage Clin. 2014 Jul 22;5:309-21. doi: 10.1016/j.nicl.2014.07.005. eCollection 2014. PMID 25161897
- [Background] Rebain R, Baxter GD, McDonough S. A systematic review of the passive straight leg raising test as a diagnostic aid for low back pain (1989 to 2000). Spine (Phila Pa 1976). 2002 Sep 1;27(17):E388-95. doi: 10.1097/00007632-200209010-00025. PMID 12221373
- [Background] Roussel NA, Nijs J, Truijen S, Smeuninx L, Stassijns G. Low back pain: clinimetric properties of the Trendelenburg test, active straight leg raise test, and breathing pattern during active straight leg raising. J Manipulative Physiol Ther. 2007 May;30(4):270-8. doi: 10.1016/j.jmpt.2007.03.001. PMID 17509436
- [Background] Skup M. Longitudinal fMRI analysis: A review of methods. Stat Interface. 2010;3(2):232-252. PMID 22655113
- [Background] Summers B, Malhan K, Cassar-Pullicino V. Low back pain on passive straight leg raising: the anterior theca as a source of pain. Spine (Phila Pa 1976). 2005 Feb 1;30(3):342-5. doi: 10.1097/01.brs.0000152378.93868.c8. PMID 15682017
- [Background] Ussher M, Cropley M, Playle S, Mohidin R, West R. Effect of isometric exercise and body scanning on cigarette cravings and withdrawal symptoms. Addiction. 2009 Jul;104(7):1251-7. doi: 10.1111/j.1360-0443.2009.02605.x. PMID 19563567
- [Background] Wasan AD, Davar G, Jamison R. The association between negative affect and opioid analgesia in patients with discogenic low back pain. Pain. 2005 Oct;117(3):450-461. doi: 10.1016/j.pain.2005.08.006. PMID 16154274
- [Background] Wasan AD, Loggia ML, Chen LQ, Napadow V, Kong J, Gollub RL. Neural correlates of chronic low back pain measured by arterial spin labeling. Anesthesiology. 2011 Aug;115(2):364-74. doi: 10.1097/ALN.0b013e318220e880. PMID 21720241
- [Background] White G (1908) Natural History and Antiquities of Selborne. London, England: Cassell and Company.
- [Background] Zeidan F, Johnson SK, Gordon NS, Goolkasian P. Effects of brief and sham mindfulness meditation on mood and cardiovascular variables. J Altern Complement Med. 2010 Aug;16(8):867-73. doi: 10.1089/acm.2009.0321. PMID 20666590
- [Background] Zeidan F, Lobanov OV, Kraft RA, Coghill RC. Brain mechanisms supporting violated expectations of pain. Pain. 2015 Sep;156(9):1772-1785. doi: 10.1097/j.pain.0000000000000231. PMID 26083664
- [Background] Zeidan F, Johnson SK, Diamond BJ, David Z, Goolkasian P. Mindfulness meditation improves cognition: evidence of brief mental training. Conscious Cogn. 2010 Jun;19(2):597-605. doi: 10.1016/j.concog.2010.03.014. Epub 2010 Apr 3. PMID 20363650
- [Background] Zeidan F, Martucci KT, Kraft RA, Gordon NS, McHaffie JG, Coghill RC. Brain mechanisms supporting the modulation of pain by mindfulness meditation. J Neurosci. 2011 Apr 6;31(14):5540-8. doi: 10.1523/JNEUROSCI.5791-10.2011. PMID 21471390
- [Background] Zeidan F, Emerson NM, Farris SR, Ray JN, Jung Y, McHaffie JG, Coghill RC. Mindfulness Meditation-Based Pain Relief Employs Different Neural Mechanisms Than Placebo and Sham Mindfulness Meditation-Induced Analgesia. J Neurosci. 2015 Nov 18;35(46):15307-25. doi: 10.1523/JNEUROSCI.2542-15.2015. PMID 26586819
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on Research Standards for Chronic Low Back Pain. Int J Ther Massage Bodywork. 2015 Sep 1;8(3):16-33. doi: 10.3822/ijtmb.v8i3.295. eCollection 2015 Sep. PMID 26388962
- [Background] Sharma HA, Gupta R, Olivero W. fMRI in patients with lumbar disc disease: a paradigm to study patients over time. J Pain Res. 2011;4:401-5. doi: 10.2147/JPR.S24393. Epub 2011 Dec 7. PMID 22247623
- [Background] Zeidan F, Gordon NS, Merchant J, Goolkasian P. The effects of brief mindfulness meditation training on experimentally induced pain. J Pain. 2010 Mar;11(3):199-209. doi: 10.1016/j.jpain.2009.07.015. Epub 2009 Oct 22. PMID 19853530
- [Background] Zeidan F, Adler-Neal AL, Wells RE, Stagnaro E, May LM, Eisenach JC, McHaffie JG, Coghill RC. Mindfulness-Meditation-Based Pain Relief Is Not Mediated by Endogenous Opioids. J Neurosci. 2016 Mar 16;36(11):3391-7. doi: 10.1523/JNEUROSCI.4328-15.2016. PMID 26985045

DOCUMENTS (1):
  • Informed Consent Form (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT03354585/ICF_000.pdf